CLINICAL TRIAL: NCT02428023
Title: B-Thalasaemia Trait and Its Possible Cardioprotective Role
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: 404 General Military Hospital, Larissa (Other)
Responsible Party: Principal Investigator, ANDREANIDIS ELIAS, Director of Cardiology Department, 404 General Military Hospital, Larissa
Other Study IDs: 404 General Military Hospital
Record Dates: First submitted 2015-04-23; First posted 2015-04-28 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Beta-Thalassemia Trait; Coronary Artery Disease
Keywords: Thalassemia; trait; coronary; stroke
MeSH Terms: conditions — Coronary Artery Disease; Thalassemia; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GrThalasaemia: estimation of IMT of the carotides arteries and calcium scoring
- GrNormal: estimation of IMT of the carotides arteries and calcium scoring

SUMMARY:
Our purpose is to investigate whether thallasaemia trait offers protection against cardiovascular events and whether this can be applied to specific characteristics of these people ( better lipid profile , better blood pressure profile) as scientific literature suggests.

DETAILED DESCRIPTION:
Thallasaemia is a major problem , especially in countries around the Mediterranean sea.On the other hand ,thallasaemia trait has been shown ,in a small number of studies , to have a possible protective role against CAD and stroke.These kind of studies have been contacted in Greece also ,and usually they enroll a small number of participants. In the study, investigators will enroll 2500 subjects who serve in military units in Thesally Greece. Firstly investigators will estimate the prevalence of thallasaemia trait in this population , as it is very high in this region and at the same time investigators will retrospectively record data from their personal files (which are annually recorded).

ELIGIBILITY:
Inclusion Criteria:

1. voluntary participation,
2. Subjects with Thalassemia treat will be confirmed of their treat by electrophoresis -

Exclusion Criteria:

-

Ages: 18 Years to 57 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 2500 subjects who serve in military units in Thessaly Greece
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Cardioprotective role of Thalassemia Treat | 1 YEAR
  Cardioprotective role of Thalassemia Treat

CONTACTS AND LOCATIONS:
Overall Officials: Elias Andreanidis, PhD, Principal Investigator — 404 General Military Hospital, Larissa
Locations (1):
- 404 Military Hospital, Larissa, Greece